CLINICAL TRIAL: NCT01053273
Title: Comparative Effectiveness of Percutaneous Adhesiolysis and Caudal Epidural Steroid Injections in Low Back and/or Lower Extremity Pain: A Randomized, Equivalence Trial
Brief Title: A Randomized, Equivalence Trial of Percutaneous Lumbar Adhesiolysis and Caudal Epidural Steroid Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pain Management Center of Paducah (Other)
Responsible Party: Principal Investigator, Laxmaiah Manchikanti, MD, Medical Director, Pain Management Center of Paducah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Protocol 27
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Low Back Pain
Keywords: Low back pain; Post lumbar laminectomy syndrome; Lumbar spinal stenosis; Local anesthetic steroid; Lumbar transforaminal epidural injection; Percutaneous epidural adhesiolysis; Caudal epidural injection
MeSH Terms: conditions — Low Back Pain; Spinal Stenosis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caudal epidural Injection (Active Comparator): Group I will receive caudal epidural injections with catheterization up to S3 with local anesthetic, steroids, and 0.9% sodium chloride solution
  Interventions: Procedure: Caudal Epidural Injection
- Percutaneous Adhesiolysis (Active Comparator): Group II will receive percutaneous adhesiolysis with targeted delivery of lidocaine, 10% hypertonic sodium chloride solution, and non-particulate betamethasone
  Interventions: Procedure: percutaneous adhesiolysis

INTERVENTIONS:
Procedure: Caudal Epidural Injection — Group I will receive caudal epidural injections with catheterization up to S3 with local anesthetic, steroids, and 0.9% sodium chloride solution
  Arms: Caudal epidural Injection
Procedure: percutaneous adhesiolysis — Group II will receive percutaneous adhesiolysis with targeted delivery of lidocaine, 10% hypertonic sodium chloride solution, and non-particulate betamethasone.
  Arms: Percutaneous Adhesiolysis

SUMMARY:
The purpose of this study is to:

* evaluate the effectiveness of percutaneous epidural adhesiolysis in managing chronic low back and/or lower extremity pain in patients without post lumbar surgery syndrome or spinal stenosis and compare with fluoroscopically directed caudal epidural steroid injections.
* evaluate and compare the adverse event profile in all groups.

DETAILED DESCRIPTION:
Recruitment is indicated in patients with chronic low back pain and/or lower extremity pain without post lumbar laminectomy syndrome or spinal stenosis, non-responsive to conservative therapy with physical therapy, chiropractic, medical therapy, and fluoroscopically directed epidural injections.

This is a single-center study performed in an interventional pain management referral center in the United States.

The study involves 120 patients assigned to one of 2 groups with 60 patients in each group.

Data management analysis includes sample size justification of 40 patients in each group with a power of 80% and a 0.05% 2-sided significance level. Statistical methodology includes chi-squared statistics, Fisher's exact test, t-test, and paired t-test with significance evaluated at P value < 0.05.

ELIGIBILITY:
Inclusion criteria:

* Patients with history of lumbar surgery of at least 6 months duration in the past
* Patients over the 18 years of age
* Patients with a history of chronic function-limiting low back pain with or without lower extremity pain of at least 6 months duration
* Patients who are competent to understand the study protocol and provide voluntary, written informed consent and participate in outcome measurements

Exclusion criteria:

* Post surgery, central spinal stenosis, and facet joints as sole pain generators
* Unstable or heavy opioid use
* Uncontrolled psychiatric disorders
* Uncontrolled medical illness
* Any conditions that could interfere with the interpretation of the outcome assessments
* Pregnant or lactating women
* Patients with a history or potential for adverse reaction(s) to local anesthetics or steroid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2014-01-27 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale (NRS), Oswestry Disability Index (ODI) | Outcomes are measured at baseline and at 3, 6, 12, 18, and 24 months post-treatment.
  duration of significant pain relief, opioid intake, and return to work

SECONDARY OUTCOMES:
Adverse event profile of side effects and complications. | Adverse events are measured at baseline and at 3, 6, 12, 18, and 24 months post-treatment, and at any time during the procedure or after the procedure the adverse events are suspected or expected.
  List and look at all side effects and complications

CONTACTS AND LOCATIONS:
Overall Officials: Laxmaiah Manchikanti, Principal Investigator — Ambulatory Surgery Center, Paducah
Locations (1):
- Pain Management Center of Paducah, Paducah, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Manchikanti L, Pampati V, Cash KA. Protocol for evaluation of the comparative effectiveness of percutaneous adhesiolysis and caudal epidural steroid injections in low back and/or lower extremity pain without post surgery syndrome or spinal stenosis. Pain Physician. 2010 Mar-Apr;13(2):E91-E110. PMID 20309389